CLINICAL TRIAL: NCT04598867
Title: A Multicenter, Randomized, Double-blind, Placebo- and Active- Controlled Study to Assess the Efficacy and Safety of CD-008-0045 in Patients With Generalized Anxiety Disorder
Brief Title: A Study to Assess the Efficacy and Safety of CD-008-0045 in Patients With Generalized Anxiety Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ChemRar Research and Development Institute, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNS-CD0080045-06
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Anxiety Disorder Generalized
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — 2-((2-morpholino)ethylthio)-5-ethoxybenzimidazole

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo- and active-controlled study to assess the efficacy and safety of CD-008-0045 in patients with GAD. The primary study objective is To assess the efficacy of CD-008-0045 at a dose 20 mg BID vs Placebo and Afobazol based on the change of the total score of the Hamilton Anxiety Rating Scale (SIGH-A) structured interview at Week 8 from baseline. Treatment response is considered the difference between group CD-008-0045 and Placebo is 5.5 points decrease of the Hamilton Anxiety Rating Scale (HARS) total score from baseline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double (Participant, Investigator) Dose blinding will be performed using Placebo. Patient will receive 2 vials labeled for study drug administration as follows: 1 capsule in the morning, and evening.
  Package numbers were assigned via IWRS. Thus, during the Study Treatment period, neither the patient nor the Investigator knew the group to which the patient was allocated. Single blinding was performed during the Placebo Run-in and Follow-up periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CD-008-0045 40 mg/day (Experimental): Patients assigned to the CD-008-0045 40 mg/day group will receive 1 capsule of CD-008-0045 (20 mg) before breakfast and before dinner for 32 weeks.
  Interventions: Drug: CD-008-0045
- Placebo (Placebo Comparator): Patients assigned to the Placebo group will receive 1 placebo capsule before breakfast, and dinner for 8 weeks.
  Interventions: Drug: Placebo
- Afobazol 30 mg/day (Active Comparator): Patients assigned to the Afobazol 30 mg/day group will receive 1 tablet of Afobazol (10 mg) before breakfast, before lunch and before dinner for 8 weeks.
  Interventions: Drug: Afobazol

INTERVENTIONS:
Drug: CD-008-0045 — CD-008-0045 20 mg capsules
  Arms: CD-008-0045 40 mg/day
Drug: Placebo — Placebo capsules
  Arms: Placebo
Drug: Afobazol — Afobazol 10 mg tabletes
  Other Names: Fabomotizole
  Arms: Afobazol 30 mg/day

SUMMARY:
This is a multicenter, randomized, double-blind, placebo- and active-controlled study to assess the efficacy and safety of CD-008-0045 in patients with generalized anxiety disorder (GAD). Each patient will participate in the study for the period of approximately 37 weeks: Screening and Run-in period: 1 week; Study Treatment period: 32 weeks; Follow-up period: 4 weeks.

DETAILED DESCRIPTION:
The study drug CD-008-0045 has a multi-targeted activity, i.e., able to inhibit adrenergic, dopamine, serotonin, and histamine receptors, thus allowing to assume its wide therapeutic potential. At Screening, the patients who meet the inclusion/exclusion criteria will be included into one-week single-blind Placebo Run-in period. At Week 0 the patients will be start double-blind Placebo and active comparator treatment period. The patients will be randomized to receive CD-008-0045 40 mg daily or Placebo or Afobazol (fabomotizole) for 8 weeks. After that, there will be an open-label treatment period for 26 weeks. The potential withdrawal syndrome will be assessed during four-week Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form;
2. Age ≥18 years old;
3. Generalized anxiety disorder diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria and International Classification of Diseases (ICD-10);
4. Scores of the Hamilton Anxiety Rating Scale (SIGH-A) structured interview at Screening and Randomization Visits (Week 0):

   * Total score ≥20;
   * Item 1 (Anxious mood) and item 2 (Tension) scores ≥2 points;
5. Condition according to the CGI-S ≥4 (moderate severity and higher) at Screening and Randomization Visits (Week 0);
6. Consent of patients to use adequate contraception methods throughout the study. Adequate contraception methods include:

   * Condoms with spermicide for males;
   * For females (at their discretion):

     * oral contraceptives,
     * condoms with spermicide (for the partner),
     * diaphragm with spermicide,
     * cervical cap with spermicide,
     * intrauterine device (IUD);
7. Ability to comply with all Study Protocol requirements;
8. 80% to 120% compliance during Run-in period, as assessed at Randomization Visit (Week 0).

Exclusion Criteria:

1. Pregnant or lactating women, or women planning to get pregnant during the clinical study; women of childbearing potential (including those without history of surgical sterilization and women with <2 years of post-menopause) not using adequate contraception methods;
2. Total score >13 of the Montgomery-Åsberg Depression Rating Scale (MADRS) structured interview.
3. Confirmed diagnosis of depressive episode, recurrent depressive disorder, bipolar affective disorder in history or at Screening;
4. Confirmed diagnosis of schizophrenia in history or at Screening;
5. Confirmed diagnosis of panic disorder in history or at Screening;
6. Phobic anxiety disorders (agoraphobia, social phobia, unspecified phobic anxiety disorder) in history or at Screening;
7. Disorders of personality or behavior in history or at Screening;
8. Post-traumatic stress disorder diagnosed within 12 months prior to Screening;
9. Eating disorders diagnosed within 12 months prior to Screening;
10. Obsessive-compulsive disorder in history or at Screening;
11. Epilepsy, seizures, head trauma with loss of consciousness, tumors, inflammatory, or demyelinating diseases of the central nervous system, stroke in history;
12. Pheochromocytoma;
13. Malignancies diagnosed within the last 5 years (except for the cured basal cell carcinoma);
14. Significant cardiovascular diseases at present or within 12 months prior to Screening, including: Chronic class III or IV heart failure (according to the New York Heart Association classification), severe arrhythmia requiring treatment with class Ia, Ib, Ic or III antiarrhythmic drugs, unstable angina, myocardial infarction, heart and coronary artery surgery, significant valvular heart disease, uncontrolled hypertension with systolic blood pressure >180 mm Hg and diastolic blood pressure >110 mm Hg, pulmonary embolism or deep vein thrombosis;
15. Nephrotic syndrome, moderate to severe chronic renal failure or significant renal impairment with Creatinine level >1.5 mg/dL in men and >1.4 mg/dL in women or glomerular filtration rate (GFR) <60 ml/min;
16. HIV, hepatitis B or C, history of cirrhosis; elevation of AST, ALT or serum Alkaline Phosphatase ≥ 2.5 times above the upper limit of normal or elevation of total bilirubin level ≥ 2 times above the upper limit of normal at Screening;
17. Significant dysfunctions of the thyroid gland in decompensation stage;
18. Anemia (hemoglobin level ≤105 g/L in females or ≤115 g/L in males); significant blood loss, or collection of at least one volumetric unit of donated blood (≥ 500 ml), or blood transfusion within 12 weeks prior to Screening;
19. Any uncontrolled concomitant somatic disease, including that with a stable treatment regimen;
20. Administration of drugs for generalized anxiety disorder,within 7 days prior to Screening and during throughout the study, including antidepressants, Pregabalin, benzodiazepines, antipsychotics;
21. Administration of Fluoxetine within 21 days prior to Screening and during throughout the study;
22. Previous administration of the study drug;
23. Known allergy, hypersensitivity or contraindications for use of CD-008-0045 and/or Afobazol;
24. Electroconvulsive therapy 3 months prior to screening;
25. Psychotherapy 3 months prior to screening and/or at the time of inclusion in the study;
26. Use of excluded drug therapy from the moment of Screening and throughout the study;
27. Administration of any study drug or participation in another clinical study within 3 months prior to Screening (except for cases when the patient was not administered the study drug during the study);
28. Addiction to tranquilizers or psychoactive substance abuse, including alcohol (history of episodic use is acceptable);
29. Inability to read or write; unwillingness to understand and comply with the Protocol procedures; non-compliance with drug dosage regimen or procedures which, in the Investigator's opinion, may affect the study results or the patient's safety and prevent the patient's participation in the study; any other concomitant diseases or severe mental disorders, which make the patient ineligible for participation in the study, limit the legal basis for Informed Consent procedure, or may affect the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in total score of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) at Week 8 from baseline. | Baseline to Week 8
  Mean change of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) score [the values from 0 to 56; the higher scores mean a worse outcome] [score]

SECONDARY OUTCOMES:
The frequency of decrease in total score of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) by 50% or more at week 8 from baseline | Baseline to Week 8
  Proportion of patients who demonstrate ≥ 50% decrease of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) [the values from 0 to 56; the higher scores mean a worse outcome] total score from baseline [% of patients]
Change in total score and sum of scores of the subscales for assessment of the mental and somatic anxiety of the Hamilton Anxiety Rating Scale (SIGH-A) structured interview for each parameter at Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32 | Baseline to Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32
  Mean change of the score sum of the mental and somatic anxiety subscales of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) [the values from 0 to 24 (the mental subscale) and from 0 to 32 (the somatic subscale); the higher scores mean a worse outcome] score [score]
Change of score of items 1 (Anxious mood) and 2 (Tension) of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) from baseline at Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32 | Baseline to Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32
  Mean change of the score in items 1 (Anxious mood) and 2 (Tension) of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) [the values from 0 to 4; the higher scores mean a worse outcome] [score]
Proportion of patients who reached a medically induced remission (the sum of scores of the SIGH-A ≤ 7) at Week 8 and Week32 | Baseline to Week 8 and Week 32
  Proportion of patients with the sum of scores of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) ≤ 7 at Week 8 and Week32
Changes in the sum of scores of the Montgomery-Asberg Depression Rating Scale (MADRS) at Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32 from baseline | Baseline to Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32
  Mean change of the Montgomery-Asberg Depression Rating Scale (MADRS) [the values from 0 to 54; the higher scores mean a worse outcome] score [score]
Change in the Clinical Global Impression-Severity (CGI-S) at Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32 from baseline | Time Frame: Baseline to Week 2, Week 2 to Week 4, Week 4 to Week 8, Week 8 to Week 16, Week 16 to Week 24, Week 24 to Week 32
  Mean change of the Clinical Global Impression-Severity (CGI-S) score [the values from 1 to 7; the higher scores mean a worse outcome] [score]
Change in the Clinical Global Impression-Improvement (CGI-I) at Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32 | Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32
  Mean change of the Clinical Global Impression-Improvement (CGI-I) score [the values from 1 to 7; the higher scores mean a worse outcome] [score]
Change of daytime somnolence level based on Visual Analogue Scale (VAS) | Baseline to Week 2, Week 4, Week 8, Week 16, Week 24 and Week 32
  Mean change of the Visual Analogue Scale (VAS) [the values from 0 to 10; the higher scores mean a worse outcome] score [score]
Change in total score of the Visual Analog Sheehan Disability Scale (SDS) at Week 8, Week 16, Week 24 and Week 32 from baseline | Baseline to Week 8, Week 16, Week 24 and Week 32
  Mean change of the Visual Analog Sheehan Disability Scale (SDS) score [the values from 0 to 10; the higher scores mean a worse outcome] [score]
Change in results of the Trail Making Test (TMT) at Week 4, Week 8, Week 16, Week 24 and Week 32 from baseline | Baseline to Week 4, Week 8, Week 16, Week 24 and Week 32
  Mean change of the Trail Making Test (TMT) results
Change in total score of the Quality of Life Scale (SF-20) at Week 8, Week 16, Week 24 and Week 32 from baseline | Baseline to Week 8, Week 16, Week 24 and Week 32
  Mean change of the Quality of Life Scale (SF-20) [the values from 0 to 78; the higher scores mean a better outcome]
Change in total score of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) at Week 4 after the last dose of therapy and baseline | Baseline to Weeks 4 after the last dose of therapy. The last dose of therapy to 4 Weeks after that
  Mean change of the Hamilton Anxiety Rating Scale structured interview (SIGH-A) [the values from 0 to 56; the higher scores mean a worse outcome] score [score]
Change in total score of the Montgomery-Asberg Depression Rating Scale (MADRS) at Week 4 after the last dose of therapy and baseline | Baseline to Weeks 4 after the last dose of therapy. The last dose of therapy to 4 Weeks after that
  Mean change of the Montgomery-Asberg Depression Rating Scale (MADRS) [the values from 0 to 54; the higher scores mean a worse outcome] score [score]
Change in the Clinical Global Impression-Severity (CGI-S) score at Week 4 after the last dose of therapy and baseline | Baseline to Weeks 4 after the last dose of therapy. The last dose of therapy to 4 Weeks after that
  Mean change of the Clinical Global Impression-Severity (CGI-S) [the values from 1 to 7; the higher scores mean a worse outcome] score [score]
Change in total score of the Visual Analog Sheehan Disability Scale (SDS) at Weeks 4 after the last dose of therapy and baseline | Baseline to Weeks 4 after the last dose of therapy. The last dose of therapy to 4 Weeks after that
  Mean change of the Visual Analog Sheehan Disability Scale (SDS) [the values from 0 to 10; the higher scores mean a worse outcome] score [score]
Change in the Clinical Global Impression-Improvement (CGI-I) at Weeks 4 after the last dose of therapy | The last dose of therapy to 4 Weeks after that
  Mean change of the Clinical Global Impression-Improvement (CGI-I) [the values from 1 to 7; the higher scores mean a worse outcome] score [score]
Concentration of CD-008-0045 and its metabolite М1 1 hour after first dose of the study drug and before next doses at visits (Ctrough) | [Time Frame: Week 4, Week 8]
  Ctrough of CD-008-0045 [ng/ml], Ctrough of M1 [ng/ml]
Impact of CYP2D6 polymorphism on the pharmacokinetic values of the study drug | [Time Frame: Week 4, Week 8]
  CYP2D6 polymorphism [type of metabolism], Ctrough of CD-008-0045 [ng/ml], Ctrough of M1 [ng/ml]

CONTACTS AND LOCATIONS:
Overall Officials: Margarita A Morozova, MD,PhD,Prof, Principal Investigator — "Research Center for Mental Health" Scientific Institution

IPD SHARING:
Plan to Share IPD: No